CLINICAL TRIAL: NCT04732780
Title: Avoidance of Hyperglycaemia in People With Type 1 Diabetes
Acronym: HYPE
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Imperial Health Charity (Other)
Responsible Party: Sponsor
Other Study IDs: 20SM6251
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Hyperglycaemia; Psychology
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire group: Individuals who attend the type 1 diabetes clinic will complete a number of self-report questionnaires and a survey.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study aims to learn more about avoidance of hyperglycaemia in adults with type 1 diabetes. People who attend a type 1 diabetes clinic will be invited to complete a number of self-report questionnaires and a survey. A subsection of people who experience avoidance of hyperglycaemia will be invited to take part in an interview in order to gain a more in-depth understanding of this issue.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes of at least 6 months duration

Exclusion Criteria:

* Inability to understand or write in the English language
* Pregnant women
* Unable to participate in the study due to other factors, as assessed by the Chief Investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with type 1 diabetes under the care of Imperial College Healthcare NHS Trust
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Oliver, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Questionnaire Group
Started | 253
Completed | 253
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Questionnaire Group
Number analyzed (Participants) | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 103
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 253

OUTCOME MEASURES:

1. Primary Outcome: Hyperglycaemia Avoidance Scale
Description: Questionnaire. Scored 0-96, with higher scores suggesting greater hyperglycaemia avoidance
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Questionnaire Group
Number analyzed (Participants) | 253
score on a scale | 44.6 (12.6)

2. Primary Outcome: General Anxiety Disorder-7 (GAD-7)
Description: Questionnaire. Scored 0-21, with higher scores suggesting greater anxiety
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Questionnaire Group
Number analyzed (Participants) | 253
score on a scale | 4 [1 to 9]

3. Primary Outcome: Patient Health Questionnaire 9 (PHQ-9)
Description: Questionnaire. Scored 0-27, with higher scores suggesting greater depression
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Questionnaire Group
Number analyzed (Participants) | 253
score on a scale | 5 [1 to 10]

4. Primary Outcome: State Trait Anxiety Inventory - Trait Subscale
Description: Questionnaire. Scored 20-80, with higher scores suggesting higher levels of trait anxiety
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Questionnaire Group
Number analyzed (Participants) | 253
score on a scale | 42.4 (12.5)

5. Primary Outcome: Hypoglycaemia Fear Survey 2 - Behaviour Subscale
Description: Questionnaire. Behaviour subscale scored 0-60; Worry subscale scored 0-72, in both cases with higher scores suggesting greater fear of hypoglycaemia.
  Please see outcome measure 7 for worry subscale results.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Questionnaire Group
Number analyzed (Participants) | 253
score on a scale | 17.2 (8.2)

6. Primary Outcome: Problem Areas in Diabetes 5
Description: Questionnaire. Scored 0-20, with higher scores suggesting greater diabetes stress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Questionnaire Group
Number analyzed (Participants) | 253
score on a scale | 8 (4.9)

7. Primary Outcome: Hypoglycaemia Fear Survey 2 - Worry Subscale
Description: Questionnaire. Behaviour subscale scored 0-60; Worry subscale scored 0-72, in both cases with higher scores suggesting greater fear of hypoglycaemia
  Please see outcome measure 5 for behaviour subscale results.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Questionnaire Group
Number analyzed (Participants) | 253
score on a scale | 26.1 (13.7)

ADVERSE EVENTS:
Time Frame: Participants spent approximately one hour completing questionnaires
Arm/Group | Questionnaire Group
All-Cause Mortality (participants affected / at risk) | 0/253
Serious Adverse Events (participants affected / at risk) | 0/253
Other Adverse Events (participants affected / at risk) | 0/253

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT04732780/Prot_SAP_000.pdf